CLINICAL TRIAL: NCT06506019
Title: Neurobiological Effects of Psilocybin in Treatment Resistant Bipolar Depression: An Emotional-Processing fMRI Pilot Study
Brief Title: Neurobiological Effects of Psilocybin in Treatment Resistant Bipolar Depression
Acronym: Psilo-BD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Joshua Rosenblat, Staff Psychiatrist, Assistant Professor, Clinician-Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-5067
Record Dates: First submitted 2024-06-26; First posted 2024-07-17 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Bipolar Depression
Keywords: Depression; Bipolar Disorder; Bipolar Depression; Treatment-Resistant Depression; Psilocybin; Psychedelics; Psychotherapy; fMRI; Bipolar Disorder II; Bipolar Disorder 2; Psilocybin-Assisted Psychotherapy
MeSH Terms: conditions — Bipolar Disorder; Depression; Depressive Disorder, Treatment-Resistant | interventions — Psilocybin; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: All participants will receive a single dose of orally administered 25mg of psilocybin taken in conjunction with supportive therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Dose Psilocybin (Experimental): Single dose of orally administered 25 mg of psilocybin taken in conjunction with supportive therapy
  Interventions: Drug: Psilocybin; Device: Functional MRI

INTERVENTIONS:
Drug: Psilocybin — 25 mg psilocybin
Device: Functional MRI — The fMRI involving resting state measures and a facial affect task will be conducted one-day and one-month after the dosing session.

SUMMARY:
This study is an open-label, single-arm, proof-of-concept study, wherein treatment resistant bipolar depression (TRBD) participants will receive one 25 mg dose of oral psilocybin accompanied by preparatory, monitoring, and integration psychotherapy sessions (psilocybin-assisted psychotherapy, or PAP). Using fMRI (functional magnetic resonance imaging), the findings of this study will provide data on the neurobiological mechanism of psilocybin in TRBD.

The primary objective is to understand the dynamic role of amygdala activity by evaluating the neurobiological effects of a single psychedelic dose (25 mg) of oral psilocybin in individuals with a moderate to severe major depressive episode and a primary diagnosis of Bipolar II Disorder, with 2 or more failed treatment trials (i.e., treatment resistant bipolar depression [TRBD]). Neurobiological effects will be determined by evaluating the association between post-treatment right amygdala activity during the facial affect task (determined by fMRI one day after the psilocybin dose) and antidepressant effects (determined by changes in the Montgomery-Åsberg Depression Rating Scale [MADRS] scores over time, during the one-week period post-psilocybin dose). This is a single-arm, open-label clinical trial wherein all participants will receive the same study intervention.

Hypothesis: Increased right amygdala activity on fMRI with emotional stimuli one day after psilocybin treatment will be associated with greater antidepressant effects in the one-week period post-treatment in individuals with TRBD.

DETAILED DESCRIPTION:
Individuals with bipolar disorder (BD) spend a third of their lives in the midst of a depressive episode. BD is a severe and persistent mental illness with a lifetime prevalence of 2-3%. Bipolar depression remains a significant treatment challenge, with a paucity of evidence-based treatments. Only four pharmacological treatments for acute bipolar depression (cariprazine, olanzapine-fluoxetine combination, quetiapine, and lurasidone) are approved by the US Food and Drug Administration (FDA). Other medications often used for the treatment of BD are those primarily used to treat mania or psychosis (i.e., lithium; antipsychotics) or major depressive disorder (MDD) (i.e., antidepressants). Lamotrigine, which is recommended by international guidelines as a maintenance treatment for BD to prevent depressive recurrence, has limited efficacy for acute BD. Current medication options are also limited by adverse effects, including renal and thyroid impairment with long-term lithium therapy and weight gain and metabolic abnormalities with atypical antipsychotics. Furthermore, treatment outcomes remain poor, particularly for depressive episodes, with over one-third of patients failing to respond to two or more first-line treatments. Hence, there is a clear need for novel and efficacious treatments for BD. However, there is a limited understanding of the neurobiology of BD, which poses as a major barrier to identifying truly innovative treatments.

Psilocybin is a chemical compound that naturally occurs in certain species of mushrooms, (for example, in the psilocybe genus, among others). It belongs to a class of drugs referred to as "psychedelics". Psilocybin is a tryptamine which is chemically similar to the neurotransmitter, serotonin, and the essential amino acid, tryptophan. It is considered a 5-hydroxytrptamineric (serotonergic) psychedelic along with other similar drugs such as dimethyltryptamine (DMT) and lysergic acid dieythamide (LSD). Psilocybin is a product for the pharmacologically active ingredient psilocin, which readily crosses the blood-brain barrier and acts as a potential partial agonist at serotonin 5HT2A and 5HT2c receptors in the brain. Typical effects of psilocybin include significantly altered states of consciousness, experienced through visual and auditory effects, changes in perception, distortions of time; and a range of effects including a sense of awe, novel perspectives, existential and personal insight, dramatically heightened empathy and feelings of compassion, strong emotions, and unitive experience. With proper screening and preparation, psilocybin has a safe physiological and psychological profile. Psilocybin is currently the preferred compound for use in clinical research involving 5-hydroxytrptaminergic psychedelics because it has a shorter duration of action and suffers from less notoriety and stigma than other similar drugs.

Two recently completed clinical trials have assessed the effects of psilocybin on TRD in participants with BDII. The first study was a non-randomized controlled trial that demonstrated a single 25 mg dose of psilocybin with accompanying PAP led to a decrease in MADRS scores in all study participants (n=15) at the 3-week primary endpoint. The second study was a randomized controlled trial that included participants with both unipolar (n=27) and bipolar treatment-resistant depression (n=4), wherein all participants received at least one 25 mg dose of psilocybin with accompanying PAP (with the exception of one participant who dropped out of the study before receiving the study intervention). Participants had the opportunity to receive up to two additional 25 mg doses of psilocybin with accompanying PAP, if they were eligible to receive a repeat dose as per the study protocol. Both trials demonstrated that 25 mg of psilocybin resulted in a decrease of depressive symptoms in participants with treatment-resistant bipolar depression, without increased incidence of manic or hypomanic symptoms.

Beyond the clinical benefits observed, psilocybin has provided several new insights into the neurobiology of depression, with dozens of additional, ongoing mechanistic studies underway. Neuroimaging studies evaluating the effects of psilocybin in treatment-resistant (unipolar) depression (TRD) have provided surprising neurobiological insights that have called into question several assumptions of mood disorders. In an open-label TRD trial evaluating the antidepressant and neurobiological effects of psilocybin, increased activity of the right amygdala was observed in response to fearful and happy faces post-treatment. Psilocybin's antidepressant effects were associated with increased right amygdala responses to negative emotional stimuli, an opposite effect to previous findings with selective serotonin reuptake inhibitors (SSRIs). Wherein SSRIs mitigate negative emotions, psilocybin might allow patients to feel, confront and work through them. These findings also suggest that neurobiological targets and mechanisms required to alleviate TRD, may be different from non-resistant depression, where SSRIs are often effective by reducing amygdala response to negative stimuli. Notably, the impact of psilocybin on amygdala function varies inter-individually depending on baseline mood state. More specifically, in healthy volunteers, psilocybin has been shown to decrease amygdala response to emotional stimuli, whereas in TRD, psilocybin was associated with increased amygdala response. Evaluating the effects of psilocybin in TRBD may improve the investigator's understanding of the neurobiology of bipolar depression by dynamically evaluating altered amygdala function and associated changes in depressive symptoms over time.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 65 years old.
2. Must be deemed to have capacity to provide informed consent;
3. Must sign and date the informed consent form;
4. Stated willingness to comply with all study procedures;
5. Ability to read and communicate in English, such that their literacy and comprehension is sufficient for understanding the consent form and study questionnaires, as evaluated by study staff obtaining consent;
6. Primary DSM-5 diagnosis of Bipolar II Disorder (BD-II) currently experiencing a Major Depressive Episode (MDE) without psychotic features as diagnosed by a mood disorder specialist and confirmed using the Mini-International Neuropsychiatric Interview (MINI);
7. Current MDE must be moderate to severe, as determined by the Hamilton Depression Rating Scale (HDRS-17) score greater than 20 with inadequate response to two or more adequate evidence-based treatment trials for bipolar depression, as per the 2018 CANMAT Bipolar Disorder Guidelines. Treatment trials are specific to current MDE rather than lifelong trials;
8. Ability to take oral medication;
9. Must be currently taking lamotrigine or planning on starting lamotrigine outside of the trial for the duration of the study, including the 1-month follow-up period, without changes in the medication;
10. Individuals who are capable of becoming pregnant: use of highly effective contraception for at least 3 months prior to screening and agreement to use such a method during study participation;
11. Individuals who are capable of fathering a child: use of condoms or other methods for the duration of study participation to ensure effective contraception with partner;
12. Individuals who are willing to taper off current medications for a minimum of 1-month prior to Baseline (V3, Day -1) and whose physician confirms that it is safe for them to do so;
13. Agreement to adhere to Lifestyle Considerations (section 4.5) throughout study duration.

Exclusion Criteria:

1. Pregnant as assessed by a urine pregnancy test at Screening (Visit 1) or individual's that intend to become pregnant during the study or are breastfeeding;
2. Treatment with another investigational drug or other intervention within 30 days of Screening (Visit 1);
3. Current symptoms of mania, hypomania or mixed features, as determined by the Young Mania Rating Scale (YMRS) score greater than 12;
4. History of mania or hypomania in the past 6 months as determined by psychiatric history;
5. Have a DSM-5 diagnosis of substance use disorder (excluding use of tobacco) within the preceding 12 months;
6. Have active suicidal ideation as determined by the C-SSRS and/or clinical interview Significant suicide risk is defined by suicidal ideation as endorsed by items 4 or 5 of the C-SSRS, OR active suicidality requiring involuntary inpatient treatment or recent suicide attempts within the past 3 months;
7. Any DSM-5 lifetime diagnosis of a schizophrenia-spectrum disorder; psychotic disorder (including but not limited to during previous mood episodes or substance-induced psychosis), bipolar I disorder, paranoid personality disorder, borderline personality disorder, or neurocognitive disorder as determined by medical history, the MINI clinical interview, and the International Personality Disorder Examination (IPDE) administered at V1;
8. Have contraindications to fMRI as determined by the MRI questionnaire;
9. Have a history of seizures;
10. Are taking anticonvulsants (with the exception of lamotrigine) or benzodiazepines (lorazepam up to 2mg/day is acceptable);
11. History of Steven-Johnson Syndrome (SJS) or suspected SJS as determined by medical history;
12. Any first-degree relative with a diagnosis of schizophrenia-spectrum disorder; psychotic disorder (unless substance-induced or due to a medical condition); or bipolar I disorder as determined by the family medical history form and discussions with the participant;
13. Presence of a relative or absolute contraindication to psilocybin, including a drug allergy, recent stroke history, uncontrolled hypertension, low or labile blood pressure, recent myocardial infarction, cardiac arrhythmic, severe coronary artery disease, or moderate to severe renal or hepatic impairment;
14. Presence of baseline prolonged QTc or Torsade de Pointes as measured by the ECG or a history of long QTc syndrome or related risk factors;
15. History of allergy to lamotrigine or psilocybin, or inability to tolerate lamotrigine during trial.
16. Participants who are unwilling or unable to take their lamotrigine (as prescribed by their most responsible physician) throughout the duration of the study, including up to the four-week post-dose visit, will be excluded from the study.
17. Use of classic psychedelic drugs (e.g., psilocybin, DMT, LSD, mescaline) within the previous 6 months of singing the informed consent form;
18. Use of intravenous or oral steroids within one week of the administration of psilocybin;
19. Use of S-Adenosyl methionine (SAM-e), 5-Hydroxytryptophan (5-HTP), L-tryptophan, and St. John's Wort one week prior to administration of psilocybin; and
20. Any other clinically significant physical illness including chronic infectious diseases or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if they take part in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of Amygdala Activity on fMRI with MADRS Score | Baseline to 1 and 4 weeks post psilocybin dosing
  Correlation between changes in the right amygdala signal activity on fMRI during negative emotional stimuli in the facial affect task before and after psilocybin dosing will be evaluated in relation to change in MADRS score.
Change in Depression Symptoms | Baseline to 4 weeks post psilocybin dosing
  Depression symptoms will be evaluated using change in Montgomery-Åsberg Depression Rating Scale (MADRS) score, a clinician-administered depression severity rating scale where higher scores indicate greater severity of depression symptoms on a scale of 0-60.
Clinical Global Impressions Scale (CGI) | Baseline to 1 week post psilocybin dosing
  Clinician judgement of illness severity and improvement on a seven-point Likert scale, ranging from "Normal, not at all depressed" to "Among the most extremely depressed patients" and "Very much improved" to "Very much worse". The CGI is evaluated on a scale from 0-30.
Study Recruitment and Retention Rates | Washout period to 4 week post psilocybin dosing
  Evaluating study feasibility based on recruitment and retention rates

SECONDARY OUTCOMES:
Self-Reported Depression Symptoms | Baseline to 4 weeks post psilocybin dosing
  Self-assessment of depression symptoms using the Quick Inventory for Depressive Symptomatology, Self-Report (QIDS-SR) where higher scores indicate greater severity on a scale of 0-42.
Self-Reported Anxiety Symptoms | Baseline to 4 weeks post psilocybin dosing
  Self-assessment of anxiety symptoms using the Generalized Anxiety Disorder 7-Item (GAD-7) where higher scores indicate greater severity on a scale from 0-21.
Subjective Functioning | Baseline to 4 weeks post psilocybin dosing
  Self-assessment of subjective function as measured by the Sheehan Disability Scale (SDS) where higher scores indicate greater severity of disability symptoms on a scale from 0-30.
Self-Reported Quality of Life | Baseline to 4 weeks post psilocybin dosing
  Self-assessment of quality of life measured by the World Health Organization-5, Well-Being Index (WHO-5) where higher scores indicate a better quality of life score on a scale from 0-25.
Self-Reported Rapid Changes in Depression Symptoms | Baseline to 4 weeks post psilocybin dosing
  Self-assessment of changes in depression symptoms in the past 72 hours (3 days) as measured by the McIntyre And Rosenblat Rapid Response Scale 14-Item (MARRRS-14). Higher scores indicate greater severity of depression symptoms in the last 72 hours on a scale from 0-63.
Self-Reported Cognitive Impairment | Baseline to 4 weeks post psilocybin dosing
  Self-assessment of cognitive impairment in the past 7 days as measured by the Perceived Deficits Questionnaire for Depression (PDQ-5-D) on a scale from 0-20.
Self-Reported Anhedonia Symptoms | Baseline to 4 weeks post psilocybin dosing
  Self-assessment of anhedonic symptoms (inability to experience pleasure or enjoy previously enjoyed activities) as measured by the Snaith Hamilton Pleasure Scale (SHAPS). Lower scores indicate greater severity of anhedonic symptoms on a scale from 1-56.

OTHER OUTCOMES:
Self-Reported Mystical Experience | Immediately post psilocybin dosing
  Self-assessment of the degree of mystical experiences following psilocybin administration using the Mystical Experience Questionnaire (MEQ). The MEQ assesses 4 empirically derived factors: mystical experiences, positive mood, transcendence of time and space and ineffability (e.g. inability to adequately describe experience in words). Responses are rated on a 6-point Likert scale ranging from 0 (none, not at all), through to 5 (extreme, more than ever before in my life).
Self-Reported Anhedonia Symptoms and Reward Thinking | Baseline to 4 weeks post psilocybin dosing
  Self-assessment of anhedonia symptoms across four domains: hobbies/past-times, food/drinks, social activities, and sensory experiences as measured by the Dimensional Anhedonia Rating Scale (DARS). Participants are asked to provide at least two of their own examples of what they find rewarding under each domain. The DARS is evaluated on a scale from 0-51 where lower scores indicate greater anhedonic symptoms.
Psychomotor Speed, Visual search, and Attention | Baseline to 4 weeks post psilocybin dosing
  The Trail Making Test B (TMT-B) requires participants to connect numbered circles with a pencil as quickly as possible in an alternating alphanumeric sequence respectively. Shorter time to complete these tests and fewer errors denotes higher performance.
Psychomotor Performance | Baseline to 4 weeks post psilocybin dosing
  The Digit Symbol Substitution Test (DSST) is a pencil and paper test of psychomotor performance. Participants will be key grid of numbers and matching symbols and are asked to fill as many empty boxes as possible with the symbol matching each number. The score is the number of correct number-symbol matches achieved in 90 seconds.
Phonemic Word Fluency | Baseline to 4 weeks post psilocybin dosing
  The FAS Verbal Fluency Test is a measure of phonemic word fluency. The number of words recited that begin with the letters 'F', 'A', and 'S' within a one-minute time frame serves as a measure of word fluency.
MATRICS Consensus Cognitive Battery Score | Baseline to 4 weeks post psilocybin dosing
  The MATRICS Consensus Cognitive Battery (MCCB) consists of 10 tests that measure outcomes across seven cognitive domains: speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, social cognition. T scores will be generated by the MCCB based on the corresponding raw data for each test.
Changes in Default Mode Network Connectivity | Baseline to 4 weeks post psilocybin dosing
  Resting state fMRI will be used to evaluate changes in connectivity within the default mode network by comparing pre- and post-psilocybin dose.
Association of Default Mode Network Connectivity with MADRS Score | Baseline to 4 weeks post psilocybin dosing
  Correlation of changes in MADRS score with changes DMN connectivity (measured using resting state fMRI) will be evaluated from baseline to 4 weeks post psilocybin dosing. The correlation is being assessed to determine if changes in DMN connectivity are associated with and can predict improvements in depression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Rosenblat, MD, MSc, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided